CLINICAL TRIAL: NCT00141115
Title: Pilot Trial of Levetiracetam in the Treatment of Alcohol Dependence With Comorbid Anxiety
Brief Title: Levetiracetam for the Treatment of Alcohol Dependence and Anxiety
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: UCB Pharma (Industry)
Responsible Party: Principal Investigator, John Mariani MD, research psychiatrist, New York State Psychiatric Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4773
Record Dates: First submitted 2005-08-31; First posted 2005-09-01 (Estimated); Results first posted 2017-09-15 (Actual); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Alcoholism; Generalized Anxiety Disorder; Panic Disorder; Social Phobia; Anxiety Disorders
Keywords: Substance-induced anxiety disorder
MeSH Terms: conditions — Alcoholism; Generalized Anxiety Disorder; Panic Disorder; Phobia, Social; Anxiety Disorders | interventions — Levetiracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Levetiracetam (Experimental): Levetiracetam 1500 mg BID
  Interventions: Drug: levetiracetam

INTERVENTIONS:
Drug: levetiracetam — Levetiracetam 1500 mg BID
  Other Names: keppra

SUMMARY:
The purpose of this study is to determine if levetiracetam is effective in treating alcohol dependence in patients with anxiety symptoms. The researchers hypothesize that individuals are unable to reduce or discontinue alcohol use because of significant anxiety, mood, and sleep disturbance symptoms that accompany reduction in alcohol use.

DETAILED DESCRIPTION:
Alcohol dependence is frequently associated with anxiety disorders. Treatment studies of individuals suffering from both alcohol dependence and anxiety have been limited. Anti-seizure medications have been used for the treatment of alcohol withdrawal for three decades. More recently, anti-seizure medications have been shown to reduce drinking and promote abstinence, and reduce drinking in abstinent alcoholics. Levetiracetam is a newer anti-seizure medication, with a structure different than that of other anti-seizure medications, that is safe and generally well tolerated. The Food and Drug Administration (FDA) has approved levetiracetam for use with other anti-seizure medications in the treatment of epilepsy in adults. The metabolism of levetiracetam is less complicated than older anti-seizure medications, which makes it easier to use and better tolerated, and it is not likely to interact with other medicines. Levetiracetam has been shown to prevent anxiety during sedative withdrawal, which is similar to alcohol withdrawal, in a laboratory study using mice. Levetiracetam also had anti-anxiety effects in laboratory study using mice. Given that other anti-seizure medications have been shown to be helpful in treating alcohol dependence, that levetiracetam is not likely to have interactions with other medications, and that in animals levetiracetam appeared to be helpful for treating a condition similar to alcohol dependence and anxiety, we believe it should be studied for the treatment of alcohol dependent patients with anxiety disorders.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between the ages of 18-65 who meet Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) criteria for alcohol dependence and a comorbid anxiety disorder, including: panic disorder, social phobia, generalized anxiety disorder, substance-induced anxiety disorder and anxiety disorder, no otherwise specified (NOS).
* Individuals capable of giving informed consent and capable of complying with study procedures.
* Individuals must have clinically significant anxiety.
* Individuals must have current average alcohol use over past 28 days with > 4 drinking days per week and >4 standard drinks/drinking day for women and > 5 standard drinks/drinking day for men.
* Women of child-bearing age will be included provided that they are not pregnant, based on the results of a blood pregnancy test done at the time of screening and agree to use a method of contraception with proven efficacy and not to become pregnant during the study. To confirm this, blood pregnancy tests will be repeated monthly. Women will be provided a full explanation of the potential dangers of pregnancy while on the study. If a woman becomes pregnant the study medication will be discontinued.
* Individual's breathalyzer reading at the time of signing consent must be < 0.04%.

Exclusion Criteria:

* Subjects with any current Axis I psychiatric disorder as defined by DSM-IV-Text Revision (DSM-IV-TR) supported by the Structured Clinical Interview for DSM-IV-TR Axis I Disorders, Research Version, Patient Edition (SCID-I/P) that in the investigator's judgment might require pharmacological intervention, with the exceptions of alcohol dependence and a comorbid anxiety disorder (panic disorder, social phobia, generalized anxiety disorder, substance-induced anxiety disorder and anxiety disorder, NOS). Current diagnoses of post-traumatic stress disorder (PTSD) or obsessive-compulsive disorder are exclusionary.
* Individuals with evidence of moderate to severe alcohol withdrawal that would require pharmacologic intervention.
* Individuals meeting DSM IV criteria for current cocaine or opioid dependence.
* Unstable physical disorders which might make participation hazardous such as uncontrolled hypertension and tachycardia (systolic blood pressure [SBP] > 150 mm Hg, diastolic blood pressure [DBP] > 90 mm Hg, or a sitting quietly heart rate [HR] > 100 bpm), acute hepatitis (patients with chronic mildly elevated transaminase levels ((2-3 x upper limit of normal) are acceptable) or poorly controlled diabetes.
* Patients currently taking prescribed psychotropic medications.
* Patients with a known sensitivity to levetiracetam.
* Individuals who have exhibited suicidal or homicidal behavior within the past two years or have current active suicidal ideation.
* Women who are pregnant or nursing.
* Individuals physiologically dependent on any other drugs (excluding nicotine, caffeine).
* Individuals with a history of a hazardous drinking behavior (e.g., driving while intoxicated convictions, violent crimes committed while intoxicated) will be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2004-03; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frances R Levin, MD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

REFERENCES:
- See also: STARS clinic website — http://www.columbiapsychiatry.org/research/clinics/stars.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Three participants were enrolled into this clinical trial at the New York State Psychiatric Insitute/Columbia University Medical Center.
Pre-assignment Details: Participants were enrolled under open-label conditions.
Period: Overall Study
Arm/Group | Levetiracetam
Started | 3
Completed | 2
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Levetiracetam
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Participants Who Reported Reductions in Alcohol Consumption
Description: Number of participants who reduced drinking during the trial
Time Frame: over 9 weeks of study or length of participation
Population: Number of participants who were drinking less at the end of the study compared to the beginning.
Measure: Count of Participants; unit: Participants
Groups:
- Levetiracetam 1500 mg Twice Daily: Levitiracetam 1500 mg administered twice daily under open-label conditions.
Arm/Group | Levetiracetam 1500 mg Twice Daily
Number analyzed (Participants) | 3
Participants | 3

2. Secondary Outcome: Percent of Drinking Days
Description: daily drinking assessed each of study participation, reported percent of drinking days for 28 days prior to study initiation compared to last 28 days of study participation-as reported on the Time line follow back
Time Frame: assessed daily, reported for baseline 28 days compared to last 28 days of study participation
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Levetiracetam
Number analyzed (Participants) | 3
percentage of days
  Baseline percent of drinking days | 67.9 (10.7)
  Last 28 days percent of drinking days | 27.6 (10.1)

ADVERSE EVENTS:
Groups:
- Levetiracetam 1500 mg Twice Daily: Levitiracetam 1500 mg administered twice daily under open label conditions.
Arm/Group | Levetiracetam 1500 mg Twice Daily
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

LIMITATIONS AND CAVEATS:
poor recruitment leading to small number of participants in the analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No